CLINICAL TRIAL: NCT07075432
Title: Comparison of the Effects of Pericapsular Nerve Block and Anterior Quadratus Lumborum Block on Spinal Anesthesia Position Pain and Postoperative Analgesia in Patients Undergoing Surgery Due to Intertrochanteric Femur Fracture
Brief Title: Preoperative and Postoperative Comparison of Two Nerve Blocks in Intertrochanteric Fracture Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, DİDEM ONK, Professor Dr., Erzincan University
Other Study IDs: ErzincanU-ANESTEZİ-DO-02
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Fracture Femur
Keywords: pericapsular nerve block; quadratus lumborum block, anterior; Pain, Postoperative; Fracture, intertrochanteric
MeSH Terms: conditions — Pain, Postoperative; Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup P-Pericapsular Nerve Block: Among the patients taken to the preoperative preparation room in the operating room, those who received routine ultrasound-guided pericapsular nerve block (PENG) following routine preoperative monitoring will be added to Group P. Pain measurement will be evaluated according to the NRS scale.
- Grup Q-Anterior Quadratus Lumborum Block: Among the patients taken to the preoperative preparation room in the operating room, those who underwent routine ultrasound-guided anterior quadratus lumborum (QLB-3) following routine preoperative monitoring will be added to Group Q. Pain measurement will be evaluated according to the NRS scale.

SUMMARY:
Patients with intertrochanteric femur fractures experience significant perioperative and postoperative pain. Perioperative pain can complicate and prolong the anesthesia process for patients undergoing spinal anesthesia, leading to complications in the procedure. Postoperative pain, in turn, prolongs hospital stays, delays recovery, and can lead to chronic postoperative pain due to high-dose opioid use for pain control.

The aim of this single-center, prospective, observational study is to compare the effects of pericapsular nerve block and anterior quadratus lumborum block on spinal anesthesia positioning pain and postoperative analgesia in patients undergoing surgery for intertrochanteric femur fractures. Our study distinguishes itself by providing scientific guidance, as there are no studies in the literature comparing the effects of these two blocks on spinal anesthesia positioning pain, spinal anesthesia success, and postoperative analgesia.

DETAILED DESCRIPTION:
A prospective observational study was planned to be conducted in the operating room of Erzincan Mengücek Gazi Training and Research Hospital. The study will be initiated after approval from the university ethics committee and written informed consent from the patients. A minimum of 64 patients aged 30-85 with elective intertrochanteric femur fractures scheduled for surgery under spinal anesthesia by the orthopedic clinic and ASA I, II, or III will be included in the study. Patients with an ASA risk score of IV or higher, those undergoing emergency surgery, those who refused the study or wished to withdraw later, those with Alzheimer's dementia delirium-like cognitive dysfunction, those with a history of local anesthetic drug toxicity, those with an infection at the block site, those with bleeding diatheses, those undergoing additional surgery or additional anesthetic procedures (general anesthesia), those with a history of chronic opioid use, and those receiving neuropathic pain medication will be excluded from the study. The study will be conducted over a 6-month period from May 19, 2025, to November 19, 2025. All patients will be informed about the study protocol and the procedures to be performed the day before surgery, and written informed consent will be obtained. Patients who are admitted to the preoperative preparation room in the operating room and who undergo routine preoperative monitoring and receive routine ultrasound-guided pericapsular nerve block (PENG) will be included in Group P, and those who undergo routine ultrasound-guided anterior quadratus lumborum block (QLB-3) will be included in Group Q. As is the routine perioperative approach, nasal oxygen will be administered at 2 L/min.

Patients will be transferred to the operating table for spinal anesthesia 30 minutes after the block. Hemodynamic data (SpO2, blood pressure, and pulse rate) will be recorded as is the routine preoperative and intraoperative process. During this process, the patient's resting pain before the block, dynamic pain before the block (leg pain at 15 degrees of elevation), resting pain at 30 minutes after the block, dynamic pain at 30 minutes after the block (leg pain at 15 degrees of elevation), and pain in the given position during spinal anesthesia will be recorded using a numerical rating scale (NRS). (The Numerical Rating Scale (NRS) is a pain score used to rate pain. During this score measurement, patients are asked to verbally state a number that corresponds to their pain, place a check mark on the number indicating their pain, or point to the number. The scale ranges from 0 to 10. 0 indicates no pain, while 10 represents the worst possible pain. Additionally, the anesthesiologist's block application times and whether spinal anesthesia was successful on the first attempt will be recorded. Patients in each group will be included in the group based on their demographic characteristics. After the procedure, patients will be admitted to the postoperative care unit as usual. Patients with an Aldrete score >9 will be transferred to the ward (The Aldrete Scoring System is a scoring system that reflects physiological recovery after anesthesia. This system examines five parameters: muscle activity, respiration, circulation, consciousness, and oxygen saturation. Each parameter is assigned a score of 0, 1, or 2, with a maximum total score of 10).

Patients' rest pain will be assessed and recorded using a numerical rating scale (NRS) at 1 hour, 4 hours, 8 hours, 12 hours, and 24 hours postoperatively. All patients will be routinely administered 50 mg dexketoprofen intravenously three times daily for postoperative analgesia. Additionally, as is routinely done for postoperative pain management in our hospital's orthopedic department, 1 mg/kg tramadol will be administered intravenously as rescue analgesia if the patient's Numerical Rating Scale (NRS) score is 4 or higher (Rescue analgesia is an additional analgesic procedure performed when pain persists despite routine analgesic treatment). Tramadol dosing intervals will be planned to be no less than 6 hours, and the maximum daily tramadol dose will not exceed 400 mg. The total number of analgesic medications (NSAIDs or opioids) used in addition to the nerve block administered for pain control within 24 hours postoperatively will be recorded. For postoperative patient monitoring, patients will be evaluated by a physician who is unaware of the type of block administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective intertrochanteric femur fracture surgery
* Patients with ASA I, II, or III risk scores
* Patients aged 30-85

Exclusion Criteria:

* Patients with an ASA risk score of IV or higher
* Patients undergoing emergency surgery
* Patients who refuse to participate in the study or wish to withdraw afterward
* Patients with cognitive dysfunction such as Alzheimer's, dementia, or delirium
* Patients with a history of local anesthetic drug toxicity
* Patients with an infection in the area where the block will be performed
* Patients with bleeding diatheses
* Patients undergoing additional surgery or additional anesthetic procedures (general anesthesia)
* Patients with a history of chronic opioid use and those receiving neuropathic pain treatment

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was calculated that a minimum of 64 patients should be included in the study. Patients between the ages of 30 and 85 who are scheduled for intertrochanteric femur fracture surgery by the orthopedics and traumatology clinic will be included in the study.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-11-19 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | 24 hours
  The numerical rating scale (NRS) is a pain score used to rate pain. Patients are asked to verbally indicate a number that matches their pain, place a check mark on the number indicating their pain, or point to the number. The scale ranges from 0 to 10. 0 indicates no pain, while 10 represents the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Üniversitesi, Erzincan, Merkez 24100, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No